CLINICAL TRIAL: NCT03449277
Title: Oral Nifedipine Versus Labetalol in Treatment of Postpartum Hypertension
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hossam Ahmed Abd Ellah (Other)
Collaborators: Assiut University (Other)
Responsible Party: Sponsor-Investigator, Hossam Ahmed Abd Ellah, Principal investigator, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1209-5934
Record Dates: First submitted 2018-02-19; First posted 2018-02-28 (Actual); Last update posted 2018-04-04 (Actual); Status verified 2018-04

CONDITIONS: Postpartum Preeclampsia
MeSH Terms: interventions — Tablets; Blood Pressure Monitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- take oral nifedipine tablets (Active Comparator): Women who take the oral tablets of nifedipine till discharge of hospital
  Interventions: Drug: Oral Tablet
- take oral labetalol tablets (Active Comparator): Women who take the oral tablets of labetalol till discharge of hospital
  Interventions: Drug: Oral Tablet

INTERVENTIONS:
Drug: Oral Tablet — oral labetalol tablets and oral nifedipine tablets
  Other Names: Monitoring blood pressure

SUMMARY:
Hypertensive disorders of pregnancy are important cause of severe morbidity, long-term disability and death among both mothers and their babies. In Africa and Asia, nearly one tenth of all maternal deaths are associated with hypertensive disorders of pregnancy research has focused on the antenatal complications' for both mother and baby and the risks and benefits of administering antihypertensive therapy prior to delivery hypertension disorders of pregnancy often persist following delivery and sometimes arise de novo postpartum one of the maternal complications of pre eclampsia is residual chronic hypertension in about 1/3 of cases elevated blood pressure is seen in 6%to 8% of all pregnancies hypertension (arterial pressure >140/90 mmhg) in pregnancy is classified into one of four conditions

1. chronic hypertension that precedes pregnancy
2. pre eclampsia and eclampsia: a systematic syndrome of elevated arterial pressure,proteinuria and other findings
3. pre eclampsia superimposed upon chronic hypertension
4. gestational hypertension or nonproteinuric hypertension of pregnancy

DETAILED DESCRIPTION:
Hypertensive disorders of pregnancy are important cause of severe morbidity, long-term disability and death among both mothers and their babies. In Africa and Asia, nearly one tenth of all maternal deaths are associated with hypertensive disorders of pregnancy research has focused on the antenatal complications' for both mother and baby and the risks and benefits of administering antihypertensive therapy prior to delivery hypertension disorders of pregnancy often persist following delivery and sometimes arise de novo postpartum one of the maternal complications of pre eclampsia is residual chronic hypertension in about 1/3 of cases elevated blood pressure is seen in 6%to 8% of all pregnancies hypertension (arterial pressure >140/90 mmhg) in pregnancy is classified into one of four conditions

1. chronic hypertension that precedes pregnancy
2. pre eclampsia and eclampsia: a systematic syndrome of elevated arterial pressure,proteinuria and other findings
3. pre eclampsia superimposed upon chronic hypertension
4. gestational hypertension or nonproteinuric hypertension of pregnancy evaluate the effectiveness, safety and acceptability of Oral nifedipine versus oral labetalol in treatment of persistent postpartum hypertension

ELIGIBILITY:
Inclusion Criteria:

* Women who have hypertension during pregnancy and persist after delivery till discharge of hospital about 2 days of monitoring the blood pressure

Exclusion Criteria:

Women with history of secondary hypertension Women with eclampsia who need intensive care unit admission and indicated other drugs rather than oral nifedipine and oral labetalol Women who have any contraindication to Nifedipine or labetalol

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-01-19 (Actual); Primary Completion 2019-02-01 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
control blood pressure | till discharge of hospital about two days
  duration,total dose to achieve blood pressure below the critical value between 140 and 150 mmHg systolic and 90-100 mmHg diastolic by monitoring of blood pressure

SECONDARY OUTCOMES:
Resolution of complications | till discharge of hospital about two days
  Measured by monitoring of blood pressure and monitoring of the complications
Improvement of hematological values | till discharge of hospital about two days
  By repeated Complete blood count
Side effects in both groups | till discharge of hospital about two days
  Monitoring if there is any side effect of any drug
Improvement of other investigations | till discharge of hospital about two days
  Monitoring by repeated urine analysis,other investigations

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Mahmoud, Prof, Study Director — Prof of ob& Gyn
Locations (1):
- Hossam Ahmed Abd Ellah, Asyut, Egypt

REFERENCES:
- [Background] WHO Recommendations for Prevention and Treatment of Pre-Eclampsia and Eclampsia. Geneva: World Health Organization; 2011. Available from http://www.ncbi.nlm.nih.gov/books/NBK140561/ PMID 23741776
- [Background] Abalos E, Duley L, Steyn DW, Henderson-Smart DJ. Antihypertensive drug therapy for mild to moderate hypertension during pregnancy. Cochrane Database Syst Rev. 2007 Jan 24;(1):CD002252. doi: 10.1002/14651858.CD002252.pub2. PMID 17253478
- [Background] Magee L, von Dadelszen P. Prevention and treatment of postpartum hypertension. Cochrane Database Syst Rev. 2013 Apr 30;2013(4):CD004351. doi: 10.1002/14651858.CD004351.pub3. PMID 23633317
- [Background] Geneva Foundation for Medical Education and Research 2017: hypertensive disorders in pregnancy
- [Background] ACOG technical bulletin. Hypertension in pregnancy. Number 219--January 1996 (replaces no. 91, February 1986). Committee on Technical Bulletins of the American College of Obstetricians and Gynecologists. Int J Gynaecol Obstet. 1996 May;53(2):175-83. No abstract available. PMID 8735301
- [Background] Lenfant C; National Education Program Working Group on High Blood Pressure in Pregnancy. Working group report on high blood pressure in pregnancy. J Clin Hypertens (Greenwich). 2001 Mar-Apr;3(2):75-88. doi: 10.1111/j.1524-6175.2001.00458.x. PMID 11416689